CLINICAL TRIAL: NCT04550858
Title: Effect of Treatment With REbamipide for Helicobacter Pylori Eradication Therapy
Brief Title: h.Pylori Ttt With Rebamipide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Mohamed Abdelrahman, director, Assiut University
Other Study IDs: ttt h.pylori with rebamipide
Record Dates: First submitted 2020-08-21; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: H.Pylori Infection
MeSH Terms: interventions — rebamipide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Rebamipide — rebamipide use for ttt of h.pylori infection

SUMMARY:
the primary aim is specially in resistant cases of H.pylori and in promotion of peptic ulcer

DETAILED DESCRIPTION:
Helicobacter pylori infection is the main cause of peptic ulcer (1, 2) Some consensus conferences have recommended triple therapy with a proton pump inhibitor (PPI) and two types of antibiotics for 7 days as first-line treatment when patients with peptic ulcer have Helicobacter pylori infection.(3, 4)This recommendation is based on the finding that patients with proven eradication of H. pylori have an extremely low rate of recurrence of peptic ulcer.(5) Although a well-controlled study found comparable rates of small gastric ulcer healing after eradication therapy alone without continuation of antiulcer treatment, relief of symptoms was significantly slower with eradication therapy alone. Moreover, the success rate of eradication therapy has decreased during the past few decades, and whether or not eradication is successful becomes clear only 2-4 weeks after treatment(6).

Patients with large gastric ulcer lesions are often not completely healed with H. pylori eradication alone (7) . Proton pump inhibitors (PPIs) have become the mainstay of maintenance therapy after eradication of H. pylori infection due to the associated effective healing and fast relief of symptoms without tachyphylaxis. However, PPI therapy has some risks, including dyspeptic symptom or rebound acid hypersecretion after cessation that may induce dependence (8,9) , drug interactions with other substrate of CYP2C19, and some kinds of respiratory or gastrointestinal infections . Also, the result of H. pylori eradication can be affected by such antisecretory drugs.(10) Rebamipide is a gastroprotective antiulcer drug that has been found to reduce the rate of recurrence of gastric ulcers without affecting H. pylori status, unlike antisecretory drugs such as PPIs and H2 receptor antagonists.6 and have a healing rate of about 90% at 8 weeks after eradication therapy (11) Rebamipide (2-(4- chlorobenzoylamino)-3-[2-(1H)-quinolinon-4-yl] propionic acid) prevents gastric ulcer formation by inhibiting neutrophil activation. Rebamipide stimulates prostaglandin generation in the gastric mucosa, resulting in stimulation of mucus secretion. Rebamipide inhibits H. pylori adhesion to the gastric epithelial cells.(12) The primary aim of study to evaluate whether rebamipide could improve success rates of anti-H. pylori treatment .

ELIGIBILITY:
Inclusion Criteria:

1. 20 years of age or older,
2. ulcer size, 5 mm or more in longest diameter,
3. single ulcer,
4. H. pylori positively.

Exclusion Criteria:

* use of medications such as PPIs, H2-receptor antagonists, other gastroprotective drugs, or nonsteroidal anti-inflammatory drugs within a week prior to the start of the trial, (2) previous eradication therapy for H. pylori, (3) acute or duodenal ulcer, (4) gastric ulcer with high risk of massive bleeding

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patient with h.pylori infection from assiut university hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-05 (Estimated); Primary Completion 2021-08-21 (Estimated); Study Completion 2021-09-21 (Estimated)

PRIMARY OUTCOMES:
Gastric ulcer healing rate in resistant cases of H. pylori resistant cases of h.pylori | 8 weeks
  healing rate of gastric ulcer defined as complete disappearance of the white coating

SECONDARY OUTCOMES:
Eradication of H. pylori | 8 weeks
  H. pylori status will be measured by culture testing and 13C-urea breath test . when both tests are negative H.pylori eradication will be considered successful